CLINICAL TRIAL: NCT00807391
Title: Transbronchial Catheter Aspiration Compared to Transbronchial Needle Aspiration in the Diagnosis of Peripheral Nodules and Masses of the Lung
Brief Title: Transbronchial Catheter Aspiration and Transbronchial Needle Aspiration in the Diagnosis of Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helios Klinik Ambrock (Other)
Responsible Party: Karl-Josef Franke, MD, Helios Klinik Ambrock
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HELIOS 2090
Record Dates: First submitted 2008-12-09; First posted 2008-12-11 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2009-08

CONDITIONS: Lung Cancer
Keywords: lung cancer; transbronchial biopsy; transbronchial catheter aspiration; transbronchial needle aspiration; peripheral pulmonary lesion; bronchoscopy
MeSH Terms: conditions — Lung Neoplasms | interventions — chaperonin cofactor A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TBCA/TBNA (Other): Under fluoroscopy first transbronchial forceps biopsy is performed, afterwards in random order transbronchial catheter aspiration(TBCA) and transbronchial needle aspiration (TBNA).
  Interventions: Procedure: TBCA, TBNA

INTERVENTIONS:
Procedure: TBCA, TBNA — One arm, in random order first transbronchial catheter aspiration and second transbronchial needle aspiration or vice verse, both techniques routinely used in the diagnosis of peripheral pulmonary lesions; the cytological specimens of TBCA and TBNA are in random order examined by two independent cytologists, all cytological specimens are afterwards examined by a third, supervising cytologist.
  Other Names: transbronchial biopsy

SUMMARY:
The aim of this study is prospectively to determine the diagnostic sensitivity of Transbronchial Catheter Aspiration (TBCA) in comparison with Transbronchial Needle Aspiration (TBNA) in the diagnosis of peripheral nodules and masses of the lung.

DETAILED DESCRIPTION:
The yield of transbronchial forceps biopsy under fluoroscopy in the diagnosis of peripheral lesion of the lung lies between 32 and 57%. Several studies prove an amelioration of success rates by addition of cytological methods such as TBNA, TBCA and bronchial brushing. Furthermore, for TBNA and TBCA a significantly higher yield was reported in comparison with transbronchial forceps biopsy. TBNA and TBCA are routinely used methods, both techniques are safe, the instruments used are certificated.

ELIGIBILITY:
Inclusion Criteria:

* informed consent prior to the procedure
* radiologically peripheral pulmonary lesions between 10 and 60 millimeters in diameter

Exclusion Criteria:

* endoscopically visible lung carcinoma
* no consent in further diagnostic procedures, when bronchoscopy fails to establish a diagnosis
* haemorrhagic syndrome; grave cardiac disease; oxygen saturation lower than 90 percent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Diagnostic sensitivity of transbronchial catheter aspiration in comparison with transbronchial needle aspiration. | one year

SECONDARY OUTCOMES:
Yield by combination of the applied techniques | one year

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Josef Franke, MD, Principal Investigator — Helios Klinik Ambrock
Locations (2):
- Germany (2):
  - Universitätsklinikum Essen, Institut für Pathologie, Essen, North Rhine-Westphalia
  - Helios Klinik Ambrock, Department of Pneumology and Critical Care Medicine, Hagen, North Rhine-Westphalia

REFERENCES:
- [Background] Franke KJ, Nilius G, Ruhle KH. [Frequency of cytological procedures in diagnostic bronchoscopy of peripheral pulmonary modules and masses]. Pneumologie. 2006 Nov;60(11):663-6. doi: 10.1055/s-2006-944263. German. PMID 17109263
- [Background] Gasparini S, Ferretti M, Secchi EB, Baldelli S, Zuccatosta L, Gusella P. Integration of transbronchial and percutaneous approach in the diagnosis of peripheral pulmonary nodules or masses. Experience with 1,027 consecutive cases. Chest. 1995 Jul;108(1):131-7. doi: 10.1378/chest.108.1.131. PMID 7606947
- [Background] Chechani V. Bronchoscopic diagnosis of solitary pulmonary nodules and lung masses in the absence of endobronchial abnormality. Chest. 1996 Mar;109(3):620-5. doi: 10.1378/chest.109.3.620. PMID 8617067
- [Background] Reichenberger F, Weber J, Tamm M, Bolliger CT, Dalquen P, Perruchoud AP, Soler M. The value of transbronchial needle aspiration in the diagnosis of peripheral pulmonary lesions. Chest. 1999 Sep;116(3):704-8. doi: 10.1378/chest.116.3.704. PMID 10492275
- [Background] Katis K, Inglesos E, Zachariadis E, Palamidas P, Paraskevopoulos I, Sideris G, Tamvakopoulou E, Apostolopoulou F, Rasidakis A. The role of transbronchial needle aspiration in the diagnosis of peripheral lung masses or nodules. Eur Respir J. 1995 Jun;8(6):963-6. PMID 7589384
- [Background] Franke KJ, Nilius G, Ruhle KH. Transbronchial catheter aspiration compared to forceps biopsy in the diagnosis of peripheral lung cancer. Eur J Med Res. 2009 Jan 28;14(1):13-7. doi: 10.1186/2047-783x-14-1-13. PMID 19258205